CLINICAL TRIAL: NCT01778530
Title: A Phase 2 Study of TRC105 in Patients With Recurrent Glioblastoma (GBM)
Brief Title: TRC105 for Recurrent Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to poor accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joohee Sul, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130048; 13-C-0048; NCT01757652 (obsolete NCT alias)
Record Dates: First submitted 2013-01-26; First posted 2013-01-29 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma; Anti-Angiogenesis; Radiotherapy; Malignant Glioma; Progression
MeSH Terms: conditions — Glioblastoma; Glioma; Disease Progression | interventions — carotuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRC105 for Recurrent Glioblastoma (Experimental)
  Interventions: Drug: TRC105

INTERVENTIONS:
Drug: TRC105 — Intravenous infusion.

SUMMARY:
Background:

- Glioblastoma is an aggressive type of brain cancer that often resists treatment. TRC105 is an experimental drug that blocks the growth of new blood vessels. It is being studied for possible use in treating different kinds of cancer. Researchers want to see if TRC105 can be used to treat glioblastoma that has not responded to standard treatments.

Objectives:

- To test the safety and effectiveness of TRC105 in adults who have glioblastoma that has not responded to standard treatments.

Eligibility:

- Individuals at least 18 years of age who have glioblastoma that has not responded to standard treatments.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Imaging studies and other tests will be used to study the tumor before the start of treatment.
* Participants will have 28-day (4-week) cycles of treatment.
* Participants will have TRC105 intravenously once a week. The first infusion will take about 4 hours. The length of time needed for the infusion may be slowly reduced if it is well tolerated.
* At the end of the first cycle (the first 4 weeks), the imaging studies will be repeated before continuing TRC105.
* Participants will take TRC105 for as long as the tumor does not grow and the side effects are not too severe. They will have imaging studies at the end of every cycle to evaluate the tumor.

DETAILED DESCRIPTION:
Background:

* TRC105 is an anti-angiogenic monoclonal antibody (mAb) that binds to CD105 (Endoglin), a transmembrane glycoprotein that is essential for angiogenesis, and expressed abundantly on activated vascular endothelial cells (ECs). CD105 is a member of the transforming growth factor-Beta (TGF-Beta) receptor superfamily, and modulates TGF-Beta signaling leading to EC proliferation and migration.
* Immunohistochemistry studies reveal that CD105 is preferentially expressed in blood vessels of tumor tissues as compared with normal mucosa. For patients with glioblastoma multiforme (GBM), increased expression of CD105 may correspond to worse survival times. Furthermore, expression of CD105 is essential for neovascularization, and is upregulated in the setting of (vascular endothelial growth factor ) VEGF inhibition.
* TRC105 binding to CD105 leads to inhibition of EC proliferation, neovascularization, and induces cell death via apoptosis. TRC105 may also mediate antibody-dependent cellular cytotoxicity (ADCC).

Objectives:

Primary

* To determine the radiographic response rate for patients with recurrent GBM treated with TRC105.
* To establish data regarding the anti-tumor activity of TRC105 in patients with GBM, as determined by progression free survival.

Secondary

* To obtain information regarding the safety of TRC105 in patients with recurrent GBM.
* To evaluate the health-related quality of life (HRQL) in patients while on treatment with TRC105.
* To examine the effect of TRC105 on vascular permeability as measured by percent change from baseline in the forward contrast transfer rate (Ktrans) of dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI).
* To examine the effect of TRC105 on vascular perfusion as measured by percent change from baseline in cerebral blood volume (CBV), cerebral blood flow (CBF), and mean transit time (MTT) of dynamic susceptibility contrast magnetic resonance imaging (DSC-MRI).
* To examine the effect of TRC105 on water diffusion as measured by percent change from baseline in apparent diffusion coefficient (ADC) and fractional anisotropy (FA) of diffusion magnetic resonance imaging (MRI).
* To examine the effect of TRC105 on tumor metabolism as measured by percent change from baseline in fludeoxyglucose F18 injection (FDG) uptake of positron emission tomography (PET) scan.
* To obtain preliminary data regarding how changes in serial FDG-PET scans and physiological MRI correlate with radiographic response rates and with progression free survival in patients treated with TRC105.

Eligibility:

-This is a phase II trial in patients with recurrent GBM who are VEGF therapy naive.

Design:

-Prior to treatment start, patients will undergo a magnetic resonance imaging (MRI) including MRI perfusion and diffusion scans, as well as an FDG-PET scan. Patients will then receive TRC105 as a single agent (weekly dose of 10 mg/kg IV). A cycle will consist of 4 weeks of therapy. At the end of the first cycle, the magnetic resonance (MR) imaging and FDG-PET scans will be repeated before continuing treatment. Patients who are clinically and neurologically stable, and who have radiographic stable or responding disease at the end of each cycle will continue treatment with TRC105. MRI perfusion and diffusion will be repeated after the completion of each cycle of therapy.

ELIGIBILITY:
* INCLUSION CRITERIA
* Patients must have histologically confirmed glioblastoma or gliosarcoma.
* Patients must have evidence for tumor progression by magnetic resonance imaging (MRI) or computed tomography (CT) scan. This scan should be performed within 14 days prior to registration and on a fixed dose of steroids for at least 5 days. If the steroid dose is increased between the date of imaging and registration a new baseline MR/CT is required. The same type of scan, ie, MRI or CT must be used throughout the period of protocol treatment for tumor measurement.
* Patients must have progressed after radiation therapy and must have an interval of greater
* Patients must have recovered from the toxic effects of prior therapy: 4 weeks from any investigational agent, 4 weeks from prior cytotoxic therapy, two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair. All toxicities from prior therapies should be resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) less than or equal to grade 1 (except for toxicities such as alopecia or vitiligo).
* Patients must be > 18 years old. Because no dosing or adverse event data are currently available on the use of TRC105 in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Karnofsky performance status > 60%
* Life expectancy of greater than 12 weeks.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes > 3,000/microliter
  * absolute neutrophil count > 1,500/microliter
  * platelets > 100,000/microliter
  * total bilirubin < 1.5 times ULN institutional upper limit of normal
  * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransaminase (ALT) serum glutamic pyruvic transaminase (SGPT) < 2.5 times institutional upper limit of normal
  * Prothrombin time (PT)/Partial thromboplastin time (PTT) < 1.5 times institutional upper limit of normal
* creatinine < 1.5 times ULN within normal institutional limits

OR

--creatinine clearance > 60 glomerular filtration rate for patients with creatinine

levels above institutional normal.

* hemoglobin of > 9grams/deciliter without transfusion support in the past 28 days

  * Patients must not have any significant medical illnesses that, in the investigators opinion, cannot be adequately controlled with appropriate therapy or would compromise the patients ability to tolerate this therapy
  * Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:
* They have recovered from the effects of surgery.
* They should have residual disease following resection of recurrent tumor.

To best assess the extent of residual disease post-operatively, a computed tomography (CT)/ magnetic resonance imaging (MRI) should be done:

no later than 96 hours in the immediate post-operative period and

* at least 4 weeks post-operatively, and
* within 14 days of registration, and
* on a steroid dosage that has been stable for at least 5 days.

If the steroid dose is increased between the date of imaging and registration, a new baseline MRI/CT is required on a stable steroid dosage for at least 5 days.

* The effects of TRC105 on the developing human fetus are unknown. For this reason and because antiangiogenic agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of TRC105 administration.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.
* A baseline 12 lead electrocardiogram (ECG) to be performed within 2 weeks of trial

EXCLUSION CRITERIA

* Patients who are receiving any other investigational agents and/or who have received an investigational agent in the prior 28 days.
* Patients may not have had prior therapy with vascular endothelial growth factor (VEGF) receptor inhibitors.
* Patients with a history of peptic ulcer disease or erosive gastritis within the past 6 months, unless treated for the condition and complete resolution has been documented by esophagogastroduodenoscopy (EGD).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TRC105.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

  * Exclude patients who have had angina, MI, symptomatic congestive heart failure (CHF), cerebral vascular accident (CVA), transient ischemic attack (TIA), arterial embolism, pulmonary embolism, deep vein thrombosis (DVT), percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG) within the last 6 months.
  * Exclude patients with cardiac arrhythmias > grade 2 in the last 28 days.
  * Exclude patients with chronic hypertension, systolic BP > 140 and/or diastolic BP > 90 despite optimal treatment.
  * Exclude human immunodeficiency virus (HIV)+ patients who have CD4 counts which are below the lower limit of normal for the institution
* Patients known to have a malignancy (other than their glioblastoma) that has required treatment in the last 12 months and/or is expected to require treatment in the next 12 months (except non-melanoma skin cancer or carcinoma in-situ in the cervix)
* Patients are not allowed to receive concurrent anti-coagulation, and may not have received thrombolytic or anticoagulant agents (except heparin or alteplase to maintain intravenous (IV) catheters) within 10 days prior to drug administration
* Serious or non-healing wound, ulcer or bone fracture
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months
* Evidence of bleeding diathesis or coagulopathy
* Patients with a history of hereditary hemorrhagic telangiectasia (HHT)
* Pregnant women are excluded from this study because TRC105 and antiangiogenic agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with TRC105, breastfeeding should be discontinued if the mother is treated with TRC105.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joohee Sul, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Yung WK, Mechtler L, Gleason MJ. Intravenous carboplatin for recurrent malignant glioma: a phase II study. J Clin Oncol. 1991 May;9(5):860-4. doi: 10.1200/JCO.1991.9.5.860. PMID 1849986
- [Background] FRANKEL SA, GERMAN WJ. Glioblastoma multiforme; review of 219 cases with regard to natural history, pathology, diagnostic methods, and treatment. J Neurosurg. 1958 Sep;15(5):489-503. doi: 10.3171/jns.1958.15.5.0489. No abstract available. PMID 13576192

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TRC105 for Recurrent Glioblastoma
Started | 2
Completed | 0
Not Completed | 2
Not completed — Progression on study | 1
Not completed — Adverse event/side effect | 1

BASELINE CHARACTERISTICS:
Arm/Group | TRC105 for Recurrent Glioblastoma
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (7.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Response Rate for Patients With Recurrent Glioblastoma Multiforme (GBM) Treated With TRC105.
Description: Response and progression will be evaluated by the Updated Response Assessment Criteria for High-Grade Gliomas developed by the Response Assessment in Neuro-Oncology Working Group (RANO). Complete response is complete disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks. Partial response is >/=50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks. Stable disease does not qualify for complete response, partial response, or progression. Progression is a >/=25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement obtained at baseline (if no decrease) or best response, on stable or increasing doses of corticosteroids,
Time Frame: 14 months
Population: This outcome measure was not met due to termination of the study for poor accrual.
Arm/Group | TRC105 for Recurrent Glioblastoma
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For details, see the adverse event module.
Time Frame: 5 months, 28 days
Measure: Number; unit: participants
Arm/Group | TRC105 for Recurrent Glioblastoma
Number analyzed (Participants) | 2
participants | 1

ADVERSE EVENTS:
Arm/Group | TRC105 for Recurrent Glioblastoma
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC105 for Recurrent Glioblastoma (N=2)
Infusion related reaction (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC105 for Recurrent Glioblastoma (N=2)
Fatigue (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Seizure (Nervous system disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No